CLINICAL TRIAL: NCT03135847
Title: Physiologically Relevant Prosthetic Limb Movement Feedback for Upper and Lower Extremity Amputees
Brief Title: Prosthetic Limb Movement Feedback for Upper and Lower Extremity Amputees
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Louis Stokes VA Medical Center (U.S. Federal Agency); University of Alberta (Other); HDT Robotics (Unknown); United States Department of Defense (U.S. Federal Agency); Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Paul Marasco, Principal Investigator, The Cleveland Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 16-140; W81XWH-15-1-0575 (Other Grant/Funding Number: Congressionally Directed Medical Research Programs)
Record Dates: First submitted 2017-04-17; First posted 2017-05-01 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2024-07

CONDITIONS: Prosthesis User; Amputation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Amputee and Able Bodied Subjects (Experimental): Map the locations in the skin or deeper muscle where limb movement perceptions occur. Use tactors (small robots providing touch and vibration) to mechanically provide sensation to the residual muscles in amputees and the intact muscles in able-bodied. The functional experiments will occur concurrently with development and application of new prosthetic socket designs to incorporate control and feedback.
  Interventions: Device: Tactor

INTERVENTIONS:
Device: Tactor — The tactor is a small robot providing touch and vibration.

SUMMARY:
To assess the functional characteristics and utility of upper and lower limb prosthetic devices (advanced bionic and current clinical standard-of-care) that incorporate physiologically relevant touch and/or movement feedback.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria are adults (18 years or over) with major limb amputation (at or above wrist or ankle).

-

Exclusion Criteria:

Exclusion criteria are any skin or pain conditions that would preclude ability to withstand pressures on their limb or to wear a prosthetic socket, or cognitive barriers precluding providing informed consent.

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2016-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Skin or tendon location | 36 months
  Locations in the skin or muscle of the residual where percepts of touch or movement occur.

SECONDARY OUTCOMES:
Sorting Task | 36 months
  Performance on a sorting task with and without tactor feedback.
Sense of Agency Questionnaire | 36 months
  Agreement with statements of agency and ownership related to perceptions of limb movement including unstructured self-reports.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Marasco, PhD, Principal Investigator — The Cleveland Clinic

IPD SHARING:
Plan to Share IPD: Yes
Significant scientific results and data will be shared. Final data sets will include information such as survey results, de-identified aggregate data of prosthetic users' abilities and functional outcomes, de-identified photographic/video. Non-proprietary/non-identifying data and findings will be disseminated in a timely manner through scientific seminars, meetings, and peer reviewed publications.
Time Frame: Data will be shared within the 4-year time frame following the end of active protocols.
Access Criteria: Data will be shared under the auspices of the principal investigator and data sharing will be done through a Cleveland Clinic issued, firewall protected FTP network server. Although the final data set will be stripped of identifiers, the possibility of deductive disclosure remains. Data/documentation will be available only under data-sharing agreements that provide for: (1) a commitment to data use only for research purposes only and non-identification of individuals; (2) a commitment to data security with using appropriate technology; and (3) a commitment to destroying/returning data after completed analyses.